CLINICAL TRIAL: NCT00157911
Title: A Double-Blind, Randomized, Multicenter, Active-Comparative, 12-Week Study to Assess the Efficacy and Safety of the Drug in Conjunction With Another Drug in Korean Patients With Primary Hypercholesterolemia
Brief Title: A Study to Evaluate Ezetimibe in Korean Patients With Primary Hypercholesterolemia (0653-042)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-042; MK0653-042; 2005_065
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholerolemia
MeSH Terms: interventions — Ezetimibe; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653; ezetimibe / Duration of Treatment: 12 weeks
Drug: Comparator: simvastatin / Duration of Treatment: 12 weeks

SUMMARY:
Patients undergo 4-week placebo lead-in and diet period, and 12-week treatment period. Clinical efficacy and safety is evaluated at weeks 4, 8 and 12. This study takes approximately 18 weeks for an individual patient to complete including post-visit at week 14.

ELIGIBILITY:
Inclusion Criteria:

* Korean males or females at least 18 years of age with hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2002-12; Primary Completion 2003-10 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
LDL-C

SECONDARY OUTCOMES:
TC, TG, HDL-C, Apolipoprotein A1, Apolipoprotein B, lipoprotein (a), LDL-C:HDL-C ratio, TC:HDL-C ratio

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Bae JW, Kim HS, Lee SC, Han KH, Jeon ES. The safety and efficacy of ezetimibe and simvastatin combination therapy in Korean patients with primary hypercholesterolemia. Korean J Med. 2005;68(5):487-497 [in Korean].